CLINICAL TRIAL: NCT03119129
Title: The Development and Evaluation of the Ho'Ouna Pono Drug Prevention
Brief Title: The Development and Evaluation of the Ho'Ouna Pono Drug Prevention Curriculum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hawaii Pacific University (Other)
Collaborators: University of Hawaii (Other); Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DA037836-01A1 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Substance-Related Disorders
Keywords: prevention; health disparities; Native Hawaiians and other Pacific Islanders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Dynamic wait-listed control group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Four middle or intermediate schools receiving the Ho'ouna Pono curriculum in Quarter 2, Academic Year (AY) 2016-2017
  Interventions: Behavioral: Ho'ouna Pono Drug Prevention Curriculum
- Cohort 2 (Experimental): Three middle or intermediate schools receiving the Ho'ouna Pono curriculum in Quarter 3, AY 2016-2017
  Interventions: Behavioral: Ho'ouna Pono Drug Prevention Curriculum
- Cohort 3 (Experimental): Three middle or intermediate schools receiving the Ho'ouna Pono curriculum in Quarter 2, AY 2017-2018
  Interventions: Behavioral: Ho'ouna Pono Drug Prevention Curriculum
- Cohort 4 (Experimental): Three middle or intermediate schools receiving the Ho'ouna Pono curriculum in Quarter 3, AY 2017-2018
  Interventions: Behavioral: Ho'ouna Pono Drug Prevention Curriculum

INTERVENTIONS:
Behavioral: Ho'ouna Pono Drug Prevention Curriculum — Ho'ouna Pono is a school-based, culturally grounded drug prevention curriculum tailored to Native Hawaiian and Pacific Islander youth on Hawai'i Island.

SUMMARY:
The purposes of this study are to complete the development of a video-enhanced, school-based drug prevention program for rural Hawaiian youth (Ho'ouna Pono) using community-based participatory research principles and practices, and to test the efficacy and adoption of the full intervention across all middle/intermediate schools on Hawai'i Island. These purposes will be accomplished through three specific aims. AIM 1 (Year 1) is to complete the Ho'ouna Pono drug prevention curriculum initially developed and validated in a NIDA-funded pilot/feasibility study (R34 DA031306). To date, five professionally filmed video vignettes depicting drug-related problem situations specific to rural Hawaiian youth and seven interactive classroom lessons have been created, implemented in randomly selected intervention schools, and preliminarily evaluated using a pre-test, post-test control group design. Aim 1 enhances and builds upon this work by producing two new video vignettes, re-editing a "Behind the Scenes" video, developing new classroom curricular components, and synthesizing the new content with the existing curriculum. AIM 2 (Years 2-3) is to evaluate the fully conceived curriculum across all middle/intermediate schools on Hawai'i Island (N = 15) using a dynamic wait-listed control group design (Brown, Wyman, Guo, & Peña, 2006). Using this design, schools will be randomly assigned to four cohorts, and cohorts will be randomly assigned to receive the curriculum at designated times staggered across the two-year evaluation period. All participating youth will be measured at six designated time points across the two-year evaluation period. Because of the staggered implementation of the curriculum, intervention effects will differ by cohort, and earlier time points will include control schools for the initial cohorts receiving the intervention. All participating youth will receive pre-tests prior to curriculum implementation and post-tests upon curriculum completion, with youth attending schools in Cohorts 1-3 receiving follow-up evaluations. AIM 3 (Year 4) is to assess community, systemic, and curricular factors related to the implementation, adoption, and sustainability of the curriculum within public middle/intermediate schools on Hawai'i Island.

The present study is the result of seven consecutive years of NIDA-funded pre-prevention and translational pilot/feasibility drug prevention research focused on rural Hawaiian youth and communities. The overall outcome of this study will be an empirically supported, culturally grounded drug prevention curriculum relevant to Native Hawaiian and Pacific Islander youth. This study addresses the lack of prevention interventions for Native Hawaiians and other Pacific Islanders (NHOPIs) and indigenous youth populations, and directly contributes to the development of an indigenous prevention science (Okamoto, Helm, et al., 2014). It has implications for informing indigenous, Pacific Islander, and rural health disparities and health equity promotion.

ELIGIBILITY:
Inclusion Criteria: Grades 6-8 in a public or public-charter middle, intermediate, or multi-level school on Hawai'i Island -

Exclusion Criteria:

-

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 486 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-04-15 (Estimated); Study Completion 2018-04-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants using drug resistance strategies as measured by the Ho'ouna Pono Survey | 30 days
  Strategies (e.g., refuse, explain, avoid, leave) used by youth to resist offers to use drugs in the home, school, or community.
Recent substance use | 30 days
  Use of alcohol, cigarettes, marijuana, and other drugs over the past month.

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Okamoto, Ph.D., Principal Investigator — Hawaii Pacific University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown CH, Wyman PA, Guo J, Pena J. Dynamic wait-listed designs for randomized trials: new designs for prevention of youth suicide. Clin Trials. 2006;3(3):259-71. doi: 10.1191/1740774506cn152oa. PMID 16895043
- [Background] Okamoto SK, Helm S, Pel S, McClain LL, Hill AP, Hayashida JK. Developing empirically based, culturally grounded drug prevention interventions for indigenous youth populations. J Behav Health Serv Res. 2014 Jan;41(1):8-19. doi: 10.1007/s11414-012-9304-0. PMID 23188485